CLINICAL TRIAL: NCT05628532
Title: Interventional Before/After Study of the Effect of the DBLG1 System With TERUMO MEDISAFE WITH Insulin Pump on Glucose Control of Patients With Type 1 Diabetes in France. The BETTER Trial
Brief Title: DBLG1 System With TERUMO MEDISAFE WITH Insulin Pump Trial
Acronym: BETTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabeloop (Industry)
Collaborators: Icadom (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCB 2022-A01901-42
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: regulation algorithm; Diabetes Treatment; Closed loop
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Interventional single-arm open-label before/after multicentric national study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of the DBLG1 system (Experimental): After a 14-day baseline period during which the patient will use a Dexcom G6 Continuous Glucose Monitoring (CGM) and his current therapy (multiple daily injection or open-loop pump), the patient will start a 42-day treatment period with the DBLG1 system followed by an optional 42-day extension period.
  Interventions: Device: Use of the DBLG1 system

INTERVENTIONS:
Device: Use of the DBLG1 system — During the treatment period, the patient will use the DBLG1 system (consisting of a DBLG1 handset with an embedded software named loop mode, a TERUMO MEDISAFE WITH patch pump and a Dexcom continuous glucose monitoring (CGM) G6). The main function of DBLG1 System is to adjust the insulin delivery at the correct time in order to maintain the patient's blood glucose in the target range and thus minimize both hypoglycaemic events and long-term complications associated with elevated average glycemia.

SUMMARY:
This study conducted in 90 adults living with type 1 diabetes is an interventional single-arm open-label before/after multicentric national study conducted as a clinical investigation according to the law EU 2017/745 art. 62.

After a 14-day baseline period during which the patient will use a Dexcom G6 Continuous Glucose Monitoring (CGM) and his current therapy (multiple daily injection or open-loop pump), the patient will start a 42-day treatment period during which he will use the DBLG1 System, a closed loop system (including a DBLG1 handset, a TERUMO MEDISAFE WITH insulin pump, in addition to his Dexcom G6 CGM). An optional 6-week extension period with treatment will be proposed to patients agreeing to pursue the use of the DBLG1 system.

The main objective is to evaluate the safety and efficacy of the DBLG1 System with a TERUMO MEDISAFE WITH insulin pump in closed-loop for 6 weeks in 90 adults with type 1 diabetes.

Data related to their glycemia, complications, usability and quality of life will be collected.

The study is completed when all patients have their "end of study" file completed in the electronic Case Report Form (eCRF).

DETAILED DESCRIPTION:
This study conducted in 90 adults living with type 1 diabetes is an interventional single-arm open-label before/after multicentric national study conducted as a clinical investigation according to the law EU 2017/745 art. 62.

The study periods are as follows:

* 2 weeks of baseline period at home will be performed. During this baseline period, all patients will use their current therapy: MDI or competitor open-loop pump. In addition to their standard treatment, all patients will receive a Dexcom G6 coupled with the DBLG1 handset used exclusively to collect the data
* Followed by a 6 weeks period of time (treatment period): Patients will be equipped with the DBLG1 System including the Medisafe With pump in closed loop mode condition
* And finally a 6 weeks optional extension period will be performed (same conditions as for treatment period)

A comparison will be made first between the 6 weeks of study closed loop and the baseline period and second between the extension closed loop and the baseline period of each patient (each patient will be his / her own control) to evaluate statistical subtlety as a secondary objective of the study. In addition, a comparison of treatment vs extension will also be performed.

Visit 1: Inclusion and start of baseline phase for a duration of 2 weeks The investigator collects the dated and signed consents of patients who meet all inclusion and non-inclusion criteria.

All subjects keep their current treatment (MDI or competitor pumps) and start their baseline phase. All subjects receive a DBLG1 handset coupled with Dexcom G6 to collect data. In each investigation center, subjects are trained by medical staff in accordance with the instructions described in IFU.

Blood HbA1c test is performed in routine between one month before the V1 visit and V1 visit. If there is no routine HbA1c sampling during this period the investigator will prescribe a study specific HbA1c blood test.

Visit 2 : V1 + 2 weeks ± 2 days : End of baseline and start of closed loop period The subject is equipped with the DBLG1 System including Medisafe with pump and trained.

The site team will ensure and confirm the capacity of the subject to daily manage his DBLG1 System and realize the device setting initialization.

The subject is asked to complete Quality of Life questionnaires (HFSII and DDS questionnaires) and DTSQs for satisfaction with his / her current treatment.

The qualified site staff review patient's glycemia control via Yourloops during the first 6 days after the beginning of treatment. An optional visit on V2 + 3 days and / or V2 + 6 days should be organized by site staff in case of any doubts regarding the system's parameters or subject's training. These visits could be performed via a phone call. All supplementary visits and related events are collected via eCRF.

Visit 3: V2 + 6 weeks ± 2 days : End of the closed loop - Start of extension (optional) The patient equipped with the DBLG1 System can continue with the 6 weeks extension phase.

The site team may optimize the device setting if necessary. The subject is asked to complete Quality of Life questionnaires (HFSII and DDS questionnaires) and DTSQs for satisfaction with the DBLG1 System

If they refuse to participate in the extension, the patients leave the study and the material is returned to the investigation site.

Visit 4: V3 + 6 weeks ± 2 days: End of study visit The subject is asked to complete Quality of Life questionnaires (HFSII and DDS questionnaires) and DTSQ for satisfaction with the closed loop DBLG1/Medisafe with Blood HbA1c test is performed

The material is returned to the investigation site

Contact by phone calls or additional visits are allowed during the study. They might be useful to discuss treatments, system parameters and adverse events

The aim of this study is to obtain CE mark for DBLG1 System based on evaluation of safety and efficacy.

The main objective is to evaluate the safety and efficacy of the DBLG1 System in closed-loop for 6 weeks. Analysis will be made between the 6 weeks treatment with closed loop vs the 2 weeks baseline

The secondary objectives of this study are to:

assess the efficacy of DBLG1 System assess the global safety of DBLG1 System assess the compliance with closed loop during treatment / extension phase assess the quality of life and satisfaction and adherence of subjects to the system

ELIGIBILITY:
Inclusion Criteria:

1. Subject who is at least 18 years old,
2. The total daily dose required must be less than 90 units (U),
3. Subject accepting to be treated with 100 U/mL rapid-acting insulin analog,
4. Type 1 diabetes treated for at least 6 months (Patients treated by manual injection with insulin pen - MDI - or by competitor open loop systems or former closed loop patients if they stopped the closed loop system > 3 months before inclusion) with a stable insulin therapy regimen for at least 15 days,
5. HbA1c ≤ 10%,
6. Subject must be affiliated to any kind of social security,
7. Living in an area covered by a GSM (Global System for Mobile Communications) network,
8. Non-isolated patient, not living alone, or having a "resource" person living nearby and having a telephone and the key of his home,
9. Must be able to speak and be literate in French,
10. Having signed the free and informed consent form

Exclusion Criteria:

1. Subject receiving a total daily dose of insulin below 8 U,
2. Subject suffering from a serious illness or undergoing treatment that might significantly impair diabetes physiology, i.e. glucose-insulin interactions, that might interfere with the medical device (for example irregular treatment by steroids),
3. Subject with severe uncorrected hearing impairment and/or severe uncorrected problems of visual acuity,
4. Subject unable to understand and perform instructions provided by Diabeloop SA,
5. Subject willing to undergo regular MRI, CT or high-frequency electric heat treatment during the study period,
6. Subject who is unwilling or unable to maintain contact with the healthcare professional,
7. Subject using a pacemaker. There is the risk of this device adversely affecting pacemakers and causing them to malfunction,
8. Subject is unable to tolerate tape adhesive around the sensor or pump placements,
9. Has any unresolved adverse skin condition in the area of sensor placement (e.g., psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection),
10. Has taken any oral, injectable, or intravenous (IV) steroids within 8 weeks from time of inclusion visit, or plans to take any oral, injectable, or IV steroids during the study,
11. Actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks,
12. Subject is using DPP-4 inhibitor, GLP-1 agonists, metformin, α-glucosidase inhibitors, thiazolidinediones and/or other SGLT2 inhibitors at time of screening,
13. Diagnosed with chronic kidney disease (glomerular filtration < 30 mL/min or Serum creatinine > 176 µmol/L),
14. Patient who has had a pancreatectomy or who has pancreatic malfunctions or pancreatic islet transplantation or pancreas transplantation,
15. Patient on dialysis,
16. Patient with impaired hepatic functions,
17. Any other physical or psychological disease, or medication likely to interfere with the conduct of the study and interpretation of the study results as judged by the investigator,
18. Pregnant woman or woman of childbearing potential in the absence of an effective method of contraception or if she does not agree to continue using contraception for the duration of the study,
19. Patient under legal protection (curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent in 70 - 180 mg/dL glycemic range | 56 days
  Impact of the use of DBLG1 system on the time spent in the target 70-180 mg/dL during the main treatment period compared to baseline, in percentage.

SECONDARY OUTCOMES:
Percentage of time spent in specific glycemic ranges | 98 days
  Impact of the use of DBLG1 system on the time spent:
  < 54 mg/dL, 54-69 mg/dL, < 70 mg/dL, 70-140 mg/dL, 70-180 mg/dL (for extension period), 181-250 mg/dL, > 250 mg/dL during the main treatment period compared to baseline, and during the extension period compared to baseline, in percentage.
Incidence of severe hypoglycemia | 98 days
  Severe hypoglycemia is defined as hypoglycemia requiring third-party intervention OR with loss of consciousness OR involving hospitalization.
  The number of episodes, the number of patients with at least one episode (and percentage) will be described per study period and overall
Incidence of severe hyperglycemia | 98 days
  Severe hyperglycemia is defined as hyperglycemia with occurrence of ketoacidosis above 3 mmol/L OR involving hospitalization. The number of episodes, the number of patients with at least one episode (and percentage) will be described per study period and overall
Number of adverse events, adverse device effects, serious adverse events, serious adverse device effects, unanticipated serious adverse device effects | 98 days
  The number of events, number of patients with at least one event (and percentage) will be described for the following type de AEs:
  Adverse Events (AEs) Serious Adverse Events (SAEs) Adverse Device Effects (ADEs) Serious adverse Device Effects (SADEs) Unanticipated Serious adverse Device Effects (USADEs) Description will be provided overall and per study periods.
Evolution of HbA1c measured by blood sampling for patients participating in extension study phase | 98 days
  Impact of the use of DBLG1 system on the evolution of HbA1c measured at baseline and after the extension period.
Glucose management indicator (GMI) | 98 days
  Impact of the use of DBLG1 system on the Glucose management indicator (GMI) during the main treatment period compared to baseline, and during the extension period compared to baseline. The formula used to calculate GMI is: GMI(%) = 3.31 + 0.02392 x [mean glucose in mg/dL].
Average sensor glucose level | 98 days
  Impact of the use of DBLG1 system on mean CGM records during the main treatment period compared to baseline, and during the extension period compared to baseline.
Variability of the glucose level | 98 days
  Impact of the use of DBLG1 system on the variability of the glucose level measured by the glycemic variation coefficient (CV) and Standard Deviation (SD) intra patient during the main treatment period compared to baseline, and during the extension period compared to baseline.
Average dose of insulin used during the entire study | 98 days
  The average sensor glucose level is calculated per patient as the average of all its CGM records over a study period.
Percentage of time spent in closed loop mode | 98 days
  For both study and extension closed loop period, the percentage of time spent with close loop mode on will be calculated as the number of CGM records under close loop over the number of possible CGM records during the period. This endpoint will be described overall and per period concerned.
Percentage of days with >75% closed loop records | 98 days
  For both study and extension closed loop period, the percentage of days with >75% closed loop records will be described as a quantitative parameter.
Diabetes Treatment Satisfaction (DTSQs) Questionnaire items | 98 days
  The 8 DTSQ questionnaire items will be described as qualitative and quantitative outcomes at baseline, treatment and extension period. The minimum and maximum scores per item are 0 and 6, respectively. The higher the score, the more satisfied the patient is with the treatment.
  The evolution in score will be compared.
Scoring of Diabetes Treatment Satisfaction (DTSQs) Questionnaire | 98 days
  The DTSQ score is the sum of the 8 questionnaire items. It has a minimum of zero and a maximum of 36. The higher the score, the more satisfied the patient is with the treatment.
  DTSQ score will be described as continuous parameters at baseline, treatment and extension period.
  The evolution in score will be compared.
Scoring of Hypoglycemia Fear Survey (HFS II) questionnaire total score | 98 days
  The Hypoglycemia Fear Survey (HFS) II questionnaire consists of 33 items. The HFS II score has a minimum of 0 and a maximum of 132. The higher the score, the more the patient fears hypoglycemia. The total score will be described as continuous parameters at baseline and at end of study. The evolution in score will be compared.
Scoring of Hypoglycemia Fear Survey (HFS II) questionnaire - Behaviour scale | 98 days
  The 15 items in Hypoglycemia Fear Survey (HFS-B) Behavior scale measure behaviors aimed at avoiding hypoglycemia and its possible negative consequences. The HFS-B score will be described as continuous parameters at baseline and at end of study. The evolution in score will be compared. The score has a minimum of 0 and a maximum of 60. The higher the score, the more the patient fears hypoglycemia.
Scoring of Hypoglycemia Fear Survey (HFS II) questionnaire - Worrieness scale | 98 days
  The 18 items in Hypoglycemia Fear Survey (HFS-W) Worriedness scale measure various aspects relating to hypoglycemic episodes that provoke anxiety. The HFS-W score will be described as continuous parameters at baseline and at end of study. The evolution in score will be compared.
  The score has a minimum of 0 and a maximum of 72. The higher the score, the more the patient fears hypoglycemia.
Scoring of Diabetes Distress Scale (DDS) | 98 days
  The 17 items of DDS will be described both as continuous and categorical variables at baseline, treatment and extension period. Each item is rated on a 6-point scale from (1) "not a problem" to (6) "a very significant problem". Average scores will be computed and described for the four critical dimensions of distress: emotional burden, regimen distress, interpersonal distress and physician distress. The minimum and maximum scores will be 1 and 6, respectively.
  The evolution in DDS average score will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Alfred PENFORNIS, Pr, Principal Investigator — CH Sud Francilien
Locations (10):
- France (10):
  - CH Sud Francilien, Corbeil-Essonnes
  - CHU Grenoble, Grenoble
  - Groupe Hospitalier La Rochelle - Ré - Aunis, La Rochelle
  - CHU Lille - Hôpital Huriez, Lille
  - Centre du diabète DIAB-eCARE - HCL, Lyon
  - Hôpital la Conception - APHM, Marseille
  - Hôpital Nord Laennec, Nantes
  - CHU Rennes Pontchaillou, Rennes
  - CHRU de Strasbourg - Hôpital Civil, Strasbourg
  - CHU Toulouse - Hôpital de Rangueil, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided